CLINICAL TRIAL: NCT04639076
Title: Study of a Personalized vs. Standard Approach to Weight Loss Recommendations
Acronym: mPWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-2003
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss Group (Active Comparator): Participants in this arm will receive a standard behavioral weight loss approach that recommends a calorie deficit based on starting weight, a standard activity minute goal progression based on baseline activity and standard behavioral weekly counseling.
  Interventions: Behavioral: Behavioral Weight Loss Program
- Personalized Behavioral Weight Loss Group (Experimental): Participants in this arm will receive a personalized weight loss approach that recommends either a low carbohydrate or low fat calorie reduced diet; personalized activity plan with either daily or weekly bout-related goals; and eating frequency of either 3 times per day or 5-6 times per day.
  Interventions: Behavioral: Personalized Behavioral Weight Loss Program

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Program — The BWL group will receive a standard weight loss intervention based on the evidence-based interventions currently being recommended for clinical practice, with general recommendations for caloric reductions based on starting weight and progressive weekly increases of physical activity (PA). Supporting behavioral lessons based on materials used in the Diabetes Prevention Program (DPP) will also be delivered. The weight loss 'prescription' will remain consistent throughout the 3 month trial. Participants will receive digital tools including a study smart phone app that incorporates diet self-monitoring, tracking of behavioral goals, behavioral lessons and resources, and integration of data from a study-provided Wi-Fi enabled scale and physical activity tracker.
  Arms: Behavioral Weight Loss Group
Behavioral: Personalized Behavioral Weight Loss Program — The PBWL group will receive a calorie goal based on measured resting energy expenditure and baseline PA. In Weeks 1-4, participants will be randomly assigned to test patterns that manipulate diet composition (low-fat or low-carbohydrate), meal frequency (3 or 5-6 meals/day), and PA goals (weekly minutes or daily minutes goals). Following this period, the optimal combination will be identified by the participant and interventionist, based on weight loss, blood glucose, hunger and ability to adhere to the prescription. This group will receive the same supporting behavioral lessons as the BWL group along with additional resources specific to their personalized prescription. The weight loss 'prescription' will vary across the 3-month trial based on response to treatment. Participants will receive the same digital tools as the BWL group with resources specific to following the prescription they are following during any given program week.
  Arms: Personalized Behavioral Weight Loss Group

SUMMARY:
The purpose of this study is to develop and test the feasibility of a behavioral weight loss intervention that uses personalized recommendations for diet and physical activity behaviors in a behavioral weight loss program and to explore factors associated with treatment adherence and response. The 12-week intervention will utilize digital tools for self-monitoring and counseling by weight management professionals. Exploratory analyses will be conducted to determine if there are genetic, metabolomic, microbiome, or psychosocial factors associated with treatment response.

DETAILED DESCRIPTION:
The primary objective of the study is to test a personalized approach for prescribing weight loss strategies in overweight adults participating in a weight loss intervention and to determine if a personalized approach can optimize weight loss compared to a standard behavioral weight loss intervention. Thus, all participants will receive a behavioral weight loss intervention delivered via remote counseling and digital tools including a smart phone app, Wi-Fi- enabled smart scale, physical activity tracker. Participants in the personalized group will also use a continuous blood glucose monitoring (CGM) device.

The differences between the two groups will be the approach used to recommend diet and physical activity changes. The study will compare a Standard Behavioral Weight Loss (BWL) approach tested in numerous previous studies and consistent with current clinical practice, to a Personalized Behavioral Weight Loss (PBWL) approach that tests a combination of diet and physical activity prescriptions to determine the best "fit" for the participant. The PWBL group will actively use CGM information during the intervention period to inform diet and activity behaviors. Participants will be randomized in a 3:1 ratio to PBWL or BWL (i.e., 30 to PBWL and 10 to BWL).

1. Behavioral Weight Loss: The BWL group will receive a standard weight loss intervention based on the evidence-based interventions currently being recommended for clinical practice, with general recommendations for caloric reductions based on starting weight and aimed at achieving a 1-2 lb. average weekly weight loss, and progressive weekly increases of physical activity. Supporting behavioral lessons adapted from materials used in the Diabetes Prevention Program, a landmark behavioral weight loss intervention, will also be delivered. The weight loss 'prescription' will remain consistent throughout the 3 month trial.
2. Personalized Behavioral Weight Loss: The PBWL group will receive a weight loss intervention that is personalized for diet and physical activity recommendations based on a testing period where various approaches to eating and physical activity that may result in differential adherence and response are tested. Calorie recommendations will be based on measured resting energy expenditure and expected activity levels and aimed at achieving a 1-2 lb. average weekly weight loss. In the initial weeks, participants will test various diet and physical activity prescriptions. Following this period, the optimal combination will be identified by the participant, in consultation with their interventionist, based on measured blood glucose, weight loss, hunger and ability to adhere to the prescription. Diet composition (percentage of calories from fat, carbohydrates, and protein) will be personalized along with meal frequency and physical activity goals. This group will receive the same supporting behavioral lessons as the BWL group along with additional resources specific to their personalized prescription. The weight loss 'prescription' will vary across the 3-month trial based on response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-50 kg/m^2
* Normal or impaired glucose as determined by HbA1c fingerstick (<6.5%)
* Own an iPhone with a data and text messaging plan
* Have home Wi-Fi access
* Have the ability to read, write, and speak English
* Not meeting the American College of Sports Medicine recommendation of 150 minutes of Moderate to Vigorous Physical Activity each week
* Ability to attend 2 in-person assessment visits at the University of North Carolina (UNC) Weight Research Program clinic (at baseline and follow-up) and participate in 12 weekly remote visits with a study interventionist via phone or video call over the 12 week intervention
* Can obtain primary care provider consent that participation is appropriate if needed

Exclusion Criteria:

* Lost more than 10 pounds in the last 6 months and kept it off
* History of weight loss surgery
* Currently participating in another physical activity or weight loss program or research study that may interfere with participation in this study
* Currently meeting exercise recommendations of 150 minutes per week of moderate-to-vigorous physical activity
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 4 months
* Planning to relocate in the next 4 months
* Cannot attend 2 in-person assessment visits at the UNC Weight Research Program clinic (at baseline and follow-up) and participate in 12 weekly remote visits with a study interventionist via phone or video call over the 12 week intervention
* Pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program, as determined by items endorsed on the Physical Activity Readiness Questionnaire (PAR-Q)
* Diagnosis of diabetes
* Taking medications to treat prediabetes
* Report taking prescription or over the counter medication with a known impact on metabolism or weight
* Current treatment for cancer
* History of clinically diagnosed eating disorder
* Diagnosis of schizophrenia or bipolar disorder
* Hospitalization for a psychiatric diagnosis within the last year
* Report a past diagnosis of or current symptoms of alcohol or substance dependence
* Unwilling or unable to wear the CGM device continuously for the duration of the study
* On dialysis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change in weight (kg) | Baseline, Month 3
  Weight will be measured in kg on a calibrated digital scale. Greater negative changes in weight from baseline to 3 months indicate greater weight loss and better outcome.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, Month 3
  BMI will be calculated using measured weight (kg) and height (m) using the formula BMI=weight (kg)/[height (m)]^2. Greater negative changes in BMI from baseline to 3 months indicate greater weight loss and better outcome.
Change in Visual Analog Score (VAS) for hunger and fullness | Baseline, Month 3
  Subjective sensations of hunger will be measured using the Visual Analogue Scale (VAS) which measures sensations that range across a continuum of values. The VAS is a horizontal line measuring exactly 100 mm in length, anchored by word descriptors (i.e., 0=Not at all hungry, 100=Extremely hungry) at each end. At baseline and Month 3, participants will be asked to complete a three item VAS by placing a mark on the line at the point they feel represents their response to the question. The 3 items and anchors are 1) How hungry did you feel over the past week (0 mm anchor = not hungry at all; 100 mm anchor = extremely hungry); 2) How full did you feel after consuming meals over the past week (0 mm anchor = not full at all; 100 mm anchor = extremely full); 3) How full in general did you feel over the past week (0 mm anchor = not full at all; 100 mm anchor = extremely full). Larger positive change numbers would indicate a greater change in perceived hunger or fullness.
Change in dietary intake (total kcals) | Baseline, Month 3
  The Automated Self-Administered 24 hour Dietary Assessment Tool (ASA-24) is a self-administered computer-automated 24-hour recall that will be administered on one weekend day and one week day per assessment period to estimate total calorie intake. Greater negative changes indicate reduced intake.
Change in dietary intake (percent kcals from carbohydrate, fat, and protein) | Baseline, Month 3
  The Automated Self-Administered 24 hour Dietary Assessment Tool (ASA-24) is a self-administered computer-automated 24-hour recall that will be administered on one weekend day and one week day per assessment period to estimate macronutrient (% calories from carbohydrate, fat and protein) composition.
Change in weekly energy expenditure in kcals | Baseline, Month 3
  The Paffenbarger questionnaire (PPAQ) assesses amount of planned and lifestyle associated physical activity performed during a typical week. The PPAQ consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants report the frequency and duration of physical activity in the past week. Scoring yields energy expenditure from physical activity per week (kcal/kg/week). Higher scores translate into greater energy expenditure per week (i.e.,better outcome). Range is 0 - no theoretical maximum.
Percent weight change | Baseline, Month 3
  Percent of baseline weight lost or gained

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez CE, Hatley KE, Polzien K, Diamond M, Tate DF. Testing a Personalized Behavioral Weight Loss Approach Using Multifactor Prescriptions and Self-Experimentation: 12-Week mHealth Pilot Randomized Controlled Trial Results. Obes Sci Pract. 2025 Feb 4;11(1):e70051. doi: 10.1002/osp4.70051. eCollection 2025 Feb. PMID 39911449